CLINICAL TRIAL: NCT03410732
Title: Activated Autologous Dendritic Cells by Autologous Tumor Cell Membrane Proteins in Treatment of Gastric Cancer
Brief Title: Dendritic Cell-based Immunotherapy in Treatment Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LanZhou University (Other)
Responsible Party: Principal Investigator, Gui Gao, Ph D, MD, MD, Ph D, LanZhou University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LAUDC 2017001
Record Dates: First submitted 2018-01-16; First posted 2018-01-25 (Actual); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Gastric Cancer
Keywords: dendritic cell; immunotherapy; tumor cell membrane proteins
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radical surgery plus activated DCs (Experimental): In 21 days after a radical surgery, activated DCs are iv infused
  Interventions: Biological: activated DCs; Procedure: radical surgery only
- Radical surgery only (Active Comparator): Radical surgery only group as a control group
  Interventions: Procedure: radical surgery only

INTERVENTIONS:
Biological: activated DCs — autologous dendritic cells are collected and enriched from 50 ml of peripheral blood, then activated by autologous tumor cell membrane proteins. Then the activated DCs are iv infused in 21 days after a radical surgery.
  Other Names: activated DCs by autologous tumor cell membrane proteins
  Arms: Radical surgery plus activated DCs
Procedure: radical surgery only — Only radical surgery is given to the control group

SUMMARY:
Study objectives are to investigate the efficacy and safety of activated autologous dendritic cells (DCs) in treatment of gastric cancer. DCs are activated by the proteins from autologous tumor cell membrane and cytokines in vitro. The efficacy endpoints include objective response, immune-cell response, recurrent rate after a radical surgery, progression-free survival and overall survival, and the safety endpoints include adverse events, laboratory tests, ECG, ECOG-PT, etc.

DETAILED DESCRIPTION:
Study objectives are to investigate the efficacy and safety of activated autologous dendritic cells (DCs) in treatment of gastric cancer. The autologous DCs are collected and enriched from peripheral blood, and then are activated by the proteins from autologous tumor cell membrane and cytokines in vitro. The efficacy endpoints include objective response, immune-cell response, recurrent rate after a radical surgery, progression-free survival and overall survival, and the safety endpoints include adverse events, laboratory tests, ECG, ECOG-PT, etc. All patients will be followed up for at least 2 years after treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent given before any trial-specific procedure is initiated
2. Male or female, at least 18 years of age at the time of informed consent
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1
4. Life expectancy >3 months assessed during Screening
5. Documented (histologically- or cytologically-proven) gastric cancer that is can be radially removed

Exclusion Criteria:

1. Non-healing wounds on any part of the body
2. Active thrombosis, or a history of deep vein thrombosis or pulmonary embolism, within 1 month prior to surgery, unless adequately treated and stable
3. Active uncontrolled bleeding or a known bleeding diathesis
4. Significant cardiovascular disease or condition, including:

   1. Congestive heart failure currently requiring therapy
   2. Class III or IV cardiovascular disease according to the New York Heart Association's (NYHA) functional criteria (25)
   3. Need for antiarrhythmic medical therapy for a ventricular arrhythmia
   4. Severe conduction disturbance (e.g., 3rd degree heart block)
   5. Unstable angina pectoris (last episode at least 6 months prior to surgery)
   6. Uncontrolled hypertension (per the Investigator's discretion)
   7. Myocardial infarction within 6 months prior to C1/D1
5. Abnormal hematologic, renal or hepatic function as defined by the following criteria:

   1. Absolute neutrophil count (ANC) <1.5 ×109/L (1500/mm3)
   2. Hemoglobin ≤9 g/dL
   3. Platelet count <75 ×109/L (75,000/mm3)
   4. Serum creatinine >1.5 × upper limit of normal (ULN) for the institution
   5. Aspartate aminotransferase (AST) >3.5 × ULN for the institution or AST >5 × ULN for the institution in case of known liver metastases
   6. Alanine aminotransferase (ALT) >3.5 × ULN for the institution or ALT >5 × ULN for the institution in case of known liver metastases
   7. Total bilirubin >1.5 × ULN for the institution
   8. Prothrombin time as assessed by International Normalized Ratio (INR) >1.5 × ULN for the institution*
   9. Partial thromboplastin time (PTT) >1.5 × ULN for the institution*
6. Any of the following within 2 weeks prior to surgery:

   1. Any serious or uncontrolled infection
   2. Any infection requiring parenteral antibiotics
   3. Unexplained fever >38.0 °C
7. Any other life-threatening illness, significant organ system dysfunction, or clinically significant laboratory abnormality, which in the opinion of the Investigator, would either compromise the patient's safety or interfere with the evaluation of the safety of the trial treatment
8. Any kind of disorder that compromises the ability of the patient to give written informed consent and/or to comply with trial procedures or is unwilling or unable to comply with trial requirements at the discretion of the Investigator
9. Breast feeding, or plans by the patient (or the patient's partner) to become pregnant during treatment or within 4 months after the end of treatment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 3 years
  Time to progression/death or censored time

SECONDARY OUTCOMES:
recurrent rate | 3 years
  the rate of cancer recurring after surgery
overall survival rate | 5 years
  time to death or censored time
immune-cells response | 3 months
  CD4/CD8 T lymphocyte percentage change
Adverse event rate | 3 months
  Adverse event rate

CONTACTS AND LOCATIONS:
Overall Officials: Yumin Li, Principal Investigator — Lanzhou University Second Hospital
Locations (1):
- Lanzhou University Second Hospital, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: Undecided
we'll update the registration system. But final data will be summarized and published in a medical journal